CLINICAL TRIAL: NCT06502613
Title: Melatonin Phase Delay May Increase Risk of Children and Adolescent Idiopathic Scoliosis.
Brief Title: Idiopathic Scoliosis New Onset and Melatonin Phase Delay in Children
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2024-08-215
Record Dates: First submitted 2024-06-28; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Scoliosis Idiopathic; Circadian Rhythm; Melatonin
Keywords: Melatonin; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Melatonin phase delay: Salivary melatonin testing shows Melatonin phase delay
- Melatonin phase nromal, controls: Salivary melatonin testing shows normal, control group

SUMMARY:
This study aimed to investigate the prevalence and clinical significance of melatonin phase delay in children with new onset and progressive idiopathic scoliosis (IS).

DETAILED DESCRIPTION:
Scoliosis is a three-dimensional (3D) structural deformity of the spine defined as a radiological lateral curvature of the spine in the coronal plane of ≥10°. The worldwide prevalence of spinal curves ranges from 0.5% to 5% in children aged 10-16 years. The aetiopathogenesis of idiopathic scoliosis includes genetic abnormalities, neuromuscular, biomechanics, bone metabolism, hormonal factors, and lifestyle explorations. However, none of these factors has been established conclusively as a direct cause of IS.

Etiological research is crucial for the treatment and prevention of idiopathic scoliosis (IS). "Melatonin deficiency" was once one of the most promising etiological hypotheses for IS. Blood melatonin deficiency and dysfunction of its signaling pathways are widely suspected to play a significant role in adolescent idiopathic scoliosis (AIS). In 1994, Machida et al were the first to discover that melatonin deficiency caused by pinealectomy could induce changes similar to idiopathic scoliosis in chickens. Bipedal mice (standing and walking on hind limbs) that underwent pinealectomy or bipedal C57BL/6 mice naturally lacking melatonin were subsequently shown to develop scoliosis as well.

However, the relationship between circulating melatonin levels and AIS in human adolescents has shown significant discrepancies among studies. Whether IS patients have a melatonin deficiency remains to be seen. While Ahuja et al found that daytime melatonin levels in AIS patients were lower than those in normal controls, most other researchers reported no significant differences in serum melatonin, urinary melatonin metabolite levels during the day and night between IS patients and controls. Goultidis et al. even found that melatonin levels in AIS patients were higher than those in the control group. Current studies only measure melatonin concentration. The impact of changes in melatonin secretion patterns on scoliosis has not yet been reported. Our cross-sectional study found that the onset and peak of melatonin secretion were both delayed in patients with scoliosis compared to the control group. The delayed melatonin secretion could be a potential cause of scoliosis.

To fill those gaps, investigators will perform a prospective, unrandomized, observational cohort study at a scoliosis center to determine the prevalence and significance of melatonin phase delay in children with IS. All subjects underwent scoliosis screening led by the Zhejiang Provincial Government. Those with a scoliometer-measured ATR > 5 degrees and a Cobb angle > 10 degrees on X-ray were diagnosed with scoliosis. Individuals with an ATR > 5 degrees but a Cobb angle < 10 degrees on X-ray, or an ATR < 5 degrees, were classified as normal. Subjects screened with the Morning and Evening Questionnaire-5 (MEQ-5), the Pediatric Sleep Questionnaire (PSQ), and the Pittsburgh Sleep Quality Index (PSQI) are used to assess circadian rhythm and sleep quality. Routine follow-up visits will be scheduled 6 months apart up to at least 36 months to assess the new onset scoliosis. Patients diagnosed with scoliosis underwent X-ray examinations, while those not diagnosed with scoliosis were uniformly screened for scoliosis in Zhejiang Province during 2024-2027

ELIGIBILITY:
Inclusion Criteria:

* Collect saliva according to standards and complete melatonin testing

  * Complete scoliometer or X-ray assess scoliosis
  * Skeletally immature (Risser Sign 0-3)
  * Age between 6 and 15
  * Patients can understand and complete the MEQ-5, PSQ, and PSQI Questionnaire at baseline and follow-up visits
  * Informed Consent Form signed by subject or the guardian

Exclusion Criteria:

-

Ages: 6 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: * Patients with scoliosis other than idiopathic, or with other musculoskeletal or neurodevelopmental conditions that might be responsible for the scoliosis
  * History of previous spine surgery or spinal injury
  * Tumor or malignant tumor in the spine and brain
  * Leg length discrepancy more than 20 mm
  * Fail to fulfill the questionnaire or refuse to attend any further evaluation
  * Plans to relocate within the next 24 months
Sampling Method: Non-Probability Sample
Enrollment: 956 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Curve Angle | Routine follow-up visits will be scheduled 6 months apart up to 36 months
  A long standard standing whole spine radiograph will be used for measuring curve size in terms of Cobb angle according to the standard Cobb method
Angle of Trunk Rotation | Routine follow-up visits will be scheduled 6 months apart up to 36 months
  In addition to spinal X-rays, a Scoliometer can also help monitor curve progression. The Scoliometer is an inclinometer that measures the asymmetries between the sides of the trunk by measuring axial rotation in degrees. Numerous studies have found a high correlation between trunk axial rotation (ATR) values and the Cobb angles.

SECONDARY OUTCOMES:
Circadian rhythm Measurements | Baseline
  circadian rhythm as assessed by Morning and Evening Questionnaire-5 (MEQ-5)
Body mass index | Routine follow-up visits will be scheduled 6 months apart up to 36 months
  Changes in height, weight and body mass index
Sleep quality | Baseline
  The Pediatric Sleep Questionnaire (PSQ) is used to assess sleep quality
Sleep quality | Baseline
  The Pittsburgh Sleep Quality Index (PSQI) is used to assess sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Aimin Wang, MD, Study Chair — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided